CLINICAL TRIAL: NCT04509206
Title: A Virtual Nutritional Education Delivered Through a Hospital Teaching Kitchen : a Proof-of-concept Study
Brief Title: Virtual Teaching Kitchen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-39597
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Cardiac Health; Metabolic Syndrome
Keywords: virtual nutritional education; teaching kitchen; food insecurity; zoom media
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Subjects will undergo four nutritional educational classes, lasting 1 hour long, conducted over a two month period. These classes will occur on zoom and subjects will be located in their home.
  Interventions: Behavioral: Nutritional education

INTERVENTIONS:
Behavioral: Nutritional education — The curriculum for the four classes include understanding MyPlate guidelines, learn basic knife skills, meal prep, and plan, home farming and no-cook cooking.

SUMMARY:
A novel way of delivering nutritional education is through experiential learning in a teaching kitchen setting. Studies have shown that patients with metabolic syndrome who underwent a series of classes that featured nutrition recommendations and cooking classes had improved cardiac health.

Boston Medical Center (BMC) serves many underserved, low-income patients and has developed an innovative strategy to combat food insecurity and its consequences. This includes a preventative food pantry, a teaching kitchen, and a rooftop farm that provides fresh produce directly to the patients. The presence of this well-established three-pronged approach places our institution in an ideal position to develop a nutritional education intervention that supports experiential learning in this high-risk population.

Given the increasing focus on providing remote experiences to minimize contact and risk of infection with Sars-COV-2, the investigators are proposing a study where patients can benefit from nutritional education virtually. Patients with food insecurity and metabolic syndrome who utilize the food pantry will be invited to an educational program conducted on zoom. The program will be run by a registered dietician and chef who will deliver education virtually. Data will be collected using surveys, phone interviews, chart review, and home monitoring to test both the feasibility of running such an intervention virtually and to explore whether attending this program improves cardiac health in patients.

ELIGIBILITY:
Inclusion Criteria:

* Users of the food pantry
* English speaking
* Must have one of following on their EPIC problem list (Diabetes mellitus, obesity, hypertension, hyperlipidemia or obstructive sleep apnea)
* Must have documented measured blood pressure, weight, height in the 12 months prior to the intervention.

Exclusion Criteria:

* Patients with advanced dementia or uncontrolled psychiatric disease
* Non-english speakers since education delivered in the pilot in English
* Uncontrolled medical illness including hypertension, recent acute coronary syndrome, active malignancy or other condition that would make the subject unable to complete the study procedures

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
recruitment rates | 12 months
  based on number of people invited to participate, number recruited and consented and number attended
retention rates | 12 months
  based on attendance at each virtual educational session
facilitators for nutritional education | 12 months
  information will be obtained through qualitative interviews
barriers to nutritional education | 12 months
  information will be obtained through qualitative interviews

SECONDARY OUTCOMES:
knowledge of healthy foods | 12 months
  through qualitative interview
change in blood pressure (BP) | baseline, up to 6 months
  Baseline BP will be extracted from medical chart. Subjects will be provided with a home BP cuff. BP measurements performed by the patient will be recorded on the BP app. The 6 month follow BP will be extracted from the medical chart if available.
change in blood glucose | baseline, up to 6 months
  Baseline blood glucose will be extracted from medical chart. Subjects will use their own glucometer to measure their blood glucose. glucose measurements performed by the patient will be recorded on the glucometer. The 6 month follow blood glucose will be extracted from the medical chart if available.
change in hemoglobin A1c | baseline, 6 months
  Baseline will be extracted from the chart and 6 month will be extracted from the chart if available
change in weight | baseline, up to 6 months
  Baseline weight will be extracted from medical chart. Subjects will be provided with a home scale. weight measurements performed by the patient will be recorded on the scale app. The 6 month follow weight will be extracted from the medical chart if available.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi M Hamburg, MD, Principal Investigator — Dept of Cardiology, BU School of Medicine
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No